CLINICAL TRIAL: NCT06243016
Title: Breaking Prolonged Sitting with High-intensity Interval Training to Improve Cognitive and Brain Health in Older Adults: a Pilot Feasibility Trial.
Brief Title: Breaking Sitting with High-intensity Interval Training for Brain Health
Acronym: HIIT2SITLess
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Northeastern University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 23938; 1R21AG080411-01A1 (NIH)
Record Dates: First submitted 2023-10-25; First posted 2024-02-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Aging
Keywords: High-intensity interval training; Sitting; Executive functions; Inhibitory control; Episodic memory; Event-related potentials; Functional connectivity
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity Interval Training (HIIT) Breaks (Active Comparator): Sitting interrupted every 30 min by 6-min HIIT bouts.
  Interventions: Behavioral: High-Intensity Interval Training (HIIT) Breaks to Sitting
- Light-Intensity Interval Training (HIIT) Breaks (Sham Comparator): Sitting interrupted every 30 min by 6-min LIIT bouts.
  Interventions: Behavioral: Light-Intensity Interval Training (LIIT) Breaks to Sitting

INTERVENTIONS:
Behavioral: High-Intensity Interval Training (HIIT) Breaks to Sitting — HIIT Breaks: a 3.5-hour sitting will be interrupted every 30 min with 6-min HIIT Breaks. During sitting participants will engage in standardized sedentary activities. Each 6-min HIIT break comprises a one-minute warm-up, followed by a 2-minute high-intensity interval, one minute rest (sitting on a cycle ergometer) followed by another 2 minutes at high intensity.
  Arms: High-Intensity Interval Training (HIIT) Breaks
Behavioral: Light-Intensity Interval Training (LIIT) Breaks to Sitting — LIIT Breaks: a 3.5-hour sitting will be interrupted every 30 min with 6-min LIIT Breaks. Each 6-min LIIT break comprises a one-minute warm-up, followed by a 2-minute light-intensity interval, one minute rest (sitting on a cycle ergometer) followed by another 2-minute light-intensity interval.
  Arms: Light-Intensity Interval Training (HIIT) Breaks

SUMMARY:
This trial will examine whether interrupting 3.5 hours of sitting every 30 min with 6 min high intensity interval training (HIIT) breaks compared to light intensity interval training (LIIT) will improve brain health in cognitively normal older adults. This trial will test the feasibility of HIIT breaks to sitting. It will also address several important but unanswered questions: (1) Does interrupting sitting with short HIIT breaks improve frontoparietal function? (2) Can interrupting sitting with HIIT breaks improve cognitive functions?

DETAILED DESCRIPTION:
The investigators are conducting an acute, single site randomized crossover trial testing two conditions lasting 3.5 hours each with a one to four-weeks washout period: (1) Interrupting sitting with 6 min of high-intensity interval training (HIIT) every 30 min, and (2) interrupting sitting with 6-min light-intensity interval training (LIIT) every 30 min. Investigators will administer the conditions in a counterbalanced order to 54 older adults (40-75 years). Brain function will be assessed using event-related brain potentials and measures of functional connectivity derived from electroencephalography. Cognitive functions will be assessed using a modified Eriksen flanker task and an antisaccade task. Investigators will measure episodic memory using a mnemonic discrimination task.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years
2. BMI <40 kg/m2
3. Sedentary (≥ 6 h/day sitting by a survey question)
4. Physically inactive adults based on the CSEP-PATH: Physical Activity and Sedentayr Behaviour Questionnaire (PASB-Q) Adult (low or medium physical activity range equivalent to less than 300 min of moderate intensity physical activity per week)
5. Capable of exercising vigorously based on the Physical Activity Readiness Questionnaire (PARQ+)
6. Has a medical clearance for maximal exercise and HIIT from a physician
7. Normotensive or participant's blood pressure is controlled
8. Intelligence quotient (IQ) ≥85
9. Fasting plasma glucose <126 mg/dL
10. Good or corrected vision and hearing
11. Right-handed
12. No significant abnormalities on the ECG during the maximal exercise test
13. No signs and symptoms that suggest an underlying cardiovascular disease as recorded during the maximal exercise test by a study physician.
14. No indications to prematurely stop the maximal exercise test as outlined by the ACSM's Guidelines for Exercise Testing and Prescription
15. Concussion if more than 12 months before the study screening.
16. History of cancer but in full remission for at least 12 months and no history of chemotherapy, signed off by the physician or an oncologist

Exclusion Criteria:

1. Physical disability or musculoskeletal disease prohibitive to vigorous exercise
2. Learning disabilities
3. Cognitive impairment (MoCA <26)
4. Type 1 or 2 diabetes
5. Neurological condition (e.g., Multiple Sclerosis, Parkinson, Dementia, Mild Cognitive Impairment)
6. Color blindness
7. Brain injury (e.g., traumatic brain injury, stroke, concussion)
8. Migraine headaches
9. Presence of other health conditions that may be exacerbated by exercise
10. History of heart disease
11. High cholesterol not controlled by medication
12. Signs and symptoms indicative of underlying cardiovascular disease
13. A chronic pulmonary disease
14. Emphysema
15. Pulmonary embolus
16. Asthma
17. History of renal disease
18. History of seizures
19. A neuropsychiatric disorder
20. Osteoporosis if it interferes with an individual's ability to exercise
21. Severe back problems
22. Severe arthritis if it interferes with an individual's ability to exercise
23. Thyroid disorder not controlled by medication
24. Polyneuropathy
25. Sleep disorders
26. Acquired immunodeficiency syndrome (AIDS)
27. Hepatitis C
28. History of long Coronavirus Disease 2019 (COVID-19)
29. History of cancer if not in full remission for at least 12 months and if a participant had the history of chemotherapy
30. Current or past smoking <12 months
31. Corticosteroid intake < 31 days before screening
32. Opioids taken < 6 months from screening
33. Anabolic androgens taken < 31 days before screening
34. A serious illness or hospitalization in the last six months
35. Currently taking medications that can affect the central nervous system (except for anxiolytics)
36. Current participation in an ongoing trial likely to influence exercise ability or cognitive function

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in task-evoked brain activity | Immediately before intervention, 2 x during the intervention (50 min and 120 min into the intervention), and immediately after the intervention
  EEG will be used to measure event-related brain potentials including the P3b-component during an inhibitory control task.

SECONDARY OUTCOMES:
Change in cognitive functions | Immediately before intervention, 2 x during the intervention (50 min and 120 min into the intervention), and immediately after the intervention
  A modified Eriksen flanker task will be used to measure inhibitory control.
Change in cognitive functions | Immediately before intervention and immediately after the intervention
  An antisaccade tasks will be used to measure inhibitory control. A mnemonic discrimination task will be used to measure episodic memory.
Change in resting stated and task evoked brain activity | Immediately before intervention and immediately after the intervention
  EEG will be used to measure functional connectivity at rest and during engagement in inhibitory control and episodic memory tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Dominika M Pindus, Ph.D., Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Derived] Pindus DM, Paluska S, So J, Wyczesany M, Ligeza TS, Sarol J, Kuang J, Quiroz FB, Shanmugam R, Syed T, Kos M, Khan N, Hillman C, Kramer A. Breaking prolonged sitting with high-intensity interval training to improve cognitive and brain health in middle-aged and older adults: a protocol for the pilot feasibility HIIT2SITLess trial. BMJ Open. 2025 May 7;15(5):e095415. doi: 10.1136/bmjopen-2024-095415. PMID 40341152